CLINICAL TRIAL: NCT02196779
Title: Laser Fluorescent Imaging of Abdominal Skin During Abdominoplasty
Status: Completed | Type: Observational
Sponsor: Swanson Center (Other)
Responsible Party: Principal Investigator, Eric Swanson, M.D., Principal Investigator, Swanson Center
Other Study IDs: Swanson 003
Record Dates: First submitted 2014-07-19; First posted 2014-07-22 (Estimated); Last update posted 2014-11-20 (Estimated); Status verified 2014-11

CONDITIONS: Abdominal Skin Redundancy
Keywords: Abdominoplasty; circulation; skin; dissection; laser; fluorescence; imaging

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients undergoing abdominoplasty: Skin circulation to abdominal flap is evaluated during surgery using laser fluorescent imaging.

SUMMARY:
Abdominoplasty is a common cosmetic operation. Some investigators believe that the risk of complications is reduced by limiting the operative dissection. However, this can compromise the quality of the result. This study was undertaken to investigate the blood supply of the abdominoplasty skin flap during surgery using laser fluorescent imaging. An imaging agent is injected and the fluorescence is recorded using a near-infrared laser. The blood supply is tested after a limited dissection and then after a traditional dissection to determine whether an extended dissection reduces the skin circulation. The study hypothesis is that there is no difference in blood supply and the traditional abdominoplasty does not compromise skin circulation.

DETAILED DESCRIPTION:
Protocol

Laser Fluorescent Imaging of Abdominal Skin During Abdominoplasty.

Background/Purpose

Abdominoplasty (tummy tuck) is a common cosmetic operation. One of the risks of surgery is delayed wound healing caused by impaired circulation to the skin. In an effort to reduce risk, some investigators1 advocate a limited-undermining technique, with preservation of the perforating blood vessels and preservation of the Scarpa fascia of the lower abdomen. However, there is no evidence that this limited-undermining technique improves blood supply compared with a traditional abdominoplasty dissection. Such a limited dissection may compromise the cosmetic result.

This study was undertaken to investigate the blood supply of the abdominal skin during the abdominoplasty procedure. By testing the circulation at two points during the dissection, and a third time after completion of the operation, data may be obtained and used to evaluate the effect of the extent of the dissection on blood supply of the skin flap.

Laser fluorescent imaging represents an objective measurement technique that has been used to quantitate blood supply in skin flaps and other tissues. It has been used for several years to monitor the vascularity of flaps used in breast reconstruction. This technique has also been used previously in patients undergoing abdominoplasty.2

Subjects

Twenty consecutive consenting adult men and women undergoing outpatient elective abdominoplasty will be investigated using laser fluorescent imaging. By testing the blood supply at three time points, the patient serves as his or her own control.

Imaging

The SPY Elite Intraoperative Perfusion Assessment System (Lifecell Corp., Branchburg, NJ) consists of a near-infrared laser that detects fluorescence. The imaging agent, indocyanine green, is absorbed at this region of the spectrum, 800-810 nm. The imaging agent is injected intravenously. Starting within 5-10 seconds of injection, the system records images of the abdomen, showing the fluorescence, which indicates blood supply. The half-life of the imaging agent is 2.5-3 minutes. The imaging agent is metabolized by the liver. The only known risk is an allergic reaction to the imaging agent. Patients with a history of an allergic reaction to iodinated contrast dyes are excluded.

Surgery

The lipoabdominoplasty technique is performed as described by Saldanha et al.1 Following this limited dissection, 3 mL (7.5 mg) of indocyanine green is injected and the abdominal image is recorded, documenting blood supply to the lower abdomen. After further dissection, another 3 mL of imaging agent is injected and the lower abdomen is re-imaged. On completion of surgery, a third injection is administered and a final image is recorded.

Null Hypothesis

A traditional abdominoplasty dissection does not compromise circulation compared with a more limited dissection technique.

Informed Consent

Patients are informed as to the nature of the study and are told that their participation is entirely voluntary and they are free to decline, and that doing so does not in any way prejudice their treatment. Patients are informed of the small risk of an allergic reaction that will be treated if it occurs.

Patient Risk

There is no patient risk apart from a very small risk of allergic reaction, which is further reduced by excluding any patient with a known allergy to iodinated contrast dye. The study does not affect patient treatment. It offers the possibility of detection of reduced skin circulation, information that can be used by the surgeon to limit the dissection if necessary and avoid tissue loss and delayed wound healing, known complications of abdominoplasty.

Sample Size

A sample of 20 patients is anticipated, treated over a period of approximately 6 months.

Disclosure

The author has no financial interest in any of the products, devices, or drugs mentioned in this article. The author has no conflicts of interest to disclose. There was no outside funding for this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing abdominoplasty

Exclusion Criteria:

* Allergy to iodinated contrast agents
* Nonconsenting patients

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult men and women undergoing abdominoplasty.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2014-07; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Skin circulation during abdominoplasty. | 6 months
  The blood supply to the skin is evaluated intraoperatively using laser fluorescent imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Swanson, M.D., Principal Investigator — Swanson Center
Locations (1):
- Swanson Center, Leawood, Kansas, United States

REFERENCES:
- [Background] Roostaeian J, Harris R, Farkas JP, Barton FE, Kenkel JM. Comparison of Limited-Undermining Lipoabdominoplasty and Traditional Abdominoplasty Using Laser Fluorescence Imaging. Aesthet Surg J. 2014 Jul;34(5):741-7. doi: 10.1177/1090820X14532286. Epub 2014 Jul 1. PMID 24809360
- [Derived] Swanson E. Comparison of Limited and Full Dissection Abdominoplasty Using Laser Fluorescence Imaging to Evaluate Perfusion of the Abdominal Skin. Plast Reconstr Surg. 2015 Jul;136(1):31e-43e. doi: 10.1097/PRS.0000000000001376. PMID 26111330